CLINICAL TRIAL: NCT00848796
Title: Do Different Heparin Brands Influence Bleeding in Coronary Surgery
Brief Title: Comparative Study of Two Brands of Heparin Already on the Market
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southlake Regional Health Centre (Other)
Responsible Party: Dr CM Peniston, Southlake Regional Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: southlake
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Heparin Leo; Hepalean; CPB Cardiopuilmonary Bypass; CABG Coronary Artery Bypass Grafting; Anticoagulation efficacy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heparin (Other): Compare two market brands of Heparin
  Interventions: Drug: Heparin Leo and Hepalean

INTERVENTIONS:
Drug: Heparin Leo and Hepalean — Dosage based on Heparin does response curve obtained from the Medtronic HMS plus
  Other Names: Heparin Leo; Hepalean

SUMMARY:
Two heparin brands have been in the market in Canada for several years. Heparin Leo from Leo Pharma and Hepalean from Organon. The former is standardized by B.P (British pharmacopeia) while the latter is standardized by U.S.P (United states pharmacopeia). Previous studies have shown Heparin Leo to have roughly a 10% less efficacy then Hepalean. It has also been demonstrated that more protamine is required to reverse Heparin Leo. It is the investigators' intention to study the post-operative effects of the two brands of heparin and whether one of the two causes less bleeding after bypass surgery.

DETAILED DESCRIPTION:
The study protocol attempts not to change the normal protocol for cardiac surgery too much.

The two different brands of heparin-Heparin Leo (Leo pharma) and Hepalean (Organon) are randomized by the float perfusionist using the program research randomizer.A 50 ml syringe is loaded with heparin for the Anesthesiologist and labelled. A 20 ml syringe is loaded with heparin and thenn labelled. It is a double blinded trial with the surgeon and anesthetist not knowing which brand heparin is being used. All cases are isolated Coronary Artery Bypass Grafting (C.A.B.G) with no concomittant conditions. The following are the patients excluded from the trial

1. RE-DO
2. COMBINATION PROCEDURE
3. VALVE REPAIR/REPLACEMENT
4. IABP-PRE/INTRA//POST-OP
5. CELL SAVER INTRA-OP
6. ANEMIA (70 g/L)/BLEEDING DISORDER eg:Jehovah's witness,hemophilia etc.
7. USE OF APROTININ
8. SMALL ADULT < 50 KG
9. AORTIC SURGERY WITH/WITHOUT CIRC ARREST
10. EMERGENT PATIENT WITH HEART FAILURE

Heparin will be administered in the trial to elevate the A.C.T-Activated clotting time to 480 s and above and the heparin level to 300u/Kg to intiate cardio-pulmonary bypass (C.P.B). Additional heparin will be given to maintain the above-mentioned levels.

The following data will be studied

* BSA
* Height
* Weight
* Diagnosis
* Procedure
* Surgeon
* Anesthetist
* Perfusionist

Pre pump Hb Pump Hb Post pump Hb

Pre pump ACT Pump ACT Post pump ACT

Projected heparin conc. Slope Protocol heparin conc Heparin time CPB time X-clamp time Heparin (initial dose) Extra heparin on pump Prime Volume RAP Volume Pump balance ml Urine output ml Average temp on CPB Phenylephrine Amt Levofed amt Creatinine AST Calculated protamine dose at the end of the case Extra protamine given Total protamine CBC after pump Total chest tube drainage in OR ml Total patient in OR time

Pre pump Post Pump Platelet INR PTT PT

Date Time NA Plavix stopped ASA stopped Heparin stopped Coumadin stopped

FFP given Total packed cells given Total platelets given Other factors given Other blood product given Ca2+ given DDAVP given

Post-op 6 hrs 12 hrs 24 hrs Chest tube drainage (ml) Chest tube removed time Hct Platelet INR PTT

ADDITIONS Packed cells Cryo Platelets Other blood product / factors

Chest reopening Yes No The reason if yes Patient transfer date- Time

Overall we are going to look at whether their is any impact on post-operative bleeding,hospital and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Coronary Artery Bypass Surgery
* Normal Hematocrit
* Normal Creatinine
* Normal Liver function

Exclusion Criteria:

* Re-do
* Combination procedure
* Valve repair/replacement
* IABP-pre/Intra/Post-op
* Cell saver intra-op
* Anemia (70 g/L)/Bleeding disorder, e.g.,: Jehovah's witness, hemophilia etc.
* Use of aprotinin
* Small adult < 50 kg
* Aortic surgery with/without circ. arrest
* Emergent patient with heart failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Chest tube drainage | 24 to 48 hrs

SECONDARY OUTCOMES:
Amount of heparin used | 1 to 7 hrs
Amount of Protamine used | 1 to 7 hrs
Measured slope with heparin/ACT titration | 1 to 7 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Peniston, MD,FRCP, Principal Investigator — Department of Cardiac surgery-S.R.H.C
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

REFERENCES:
- [Result] Dyck L, Friesen RM. Do different heparin brands influence activated clotting times? J Extra Corpor Technol. 1998 Jun;30(2):73-6. PMID 10182116